CLINICAL TRIAL: NCT01546389
Title: A Phase I, Randomized Malaria Challenge Study of Intradermally-Administered Infectious (Replication-intact), Cryopreserved Plasmodium Falciparum Sporozoites (PfSPZ Challenge) in Malaria-Naïve Adults
Brief Title: Sanaria™ PfSPZ Challenge Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 11-0027; N01AI80057C
Record Dates: First submitted 2011-12-29; First posted 2012-03-07 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Malaria
Keywords: Malaria, vaccine, PfSPZ, challenge
MeSH Terms: conditions — Malaria | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Cohort 3, Group E (Experimental): Cohort 3 (High Dose, Low Aliquot), Group e: 50,000 PfSPZ in 2 divided doses (e.g., 25,000 PfSPZ per 10 mcL dose); 5 subjects
  Interventions: Biological: Sanaria™ PfSPZ Vaccine; Drug: Chloroquine
- Cohort 1, Group A (Experimental): Cohort 1 (Medium Dose, Medium Aliquot), Group a: 10,000 PfSPZ in 2 divided doses (e.g., 5000 PfSPZ per 50 microliter (mcL) dose); 5 subjects.
  Interventions: Biological: Sanaria™ PfSPZ Vaccine; Drug: Chloroquine
- Cohort 1, Group B (Experimental): Cohort 1 (Medium Dose, Medium Aliquot), Group b: 10,000 PfSPZ in 8 divided doses (e.g., 1250 PfSPZ per 50 mcL dose); 5 subjects
  Interventions: Biological: Sanaria™ PfSPZ Vaccine; Drug: Chloroquine
- Cohort 3, Group F (Experimental): Cohort 3 (High Dose, Low Aliquot), Group f: 50,000 PfSPZ in 8 divided doses (e.g., 6,250 PfSPZ per 10 mcL dose); 5 subjects
  Interventions: Biological: Sanaria™ PfSPZ Vaccine; Drug: Chloroquine
- Cohort 2, Group D (Experimental): Cohort 2 (Medium Dose, Low Aliquot), Group d: 10,000 PfSPZ in 8 divided doses (e.g., 1250 PfSPZ per 10 mcL dose); 5 subjects
  Interventions: Biological: Sanaria™ PfSPZ Vaccine; Drug: Chloroquine
- Cohort 2, Group C (Experimental): Cohort 2 (Medium Dose, Low Aliquot), Group c: 10,000 PfSPZ in 2 divided doses (e.g., 5000 PfSPZ per 10 mcL dose); 5 subjects
  Interventions: Biological: Sanaria™ PfSPZ Vaccine; Drug: Chloroquine

INTERVENTIONS:
Biological: Sanaria™ PfSPZ Vaccine — 30 subjects in 3 cohorts, 6 groups in different doses of PfSPZ vaccine via the intradermal route. Cohort 1 Medium Dose, Medium Aliquot: Group a: 10,000 PfSPZ in 2 divided doses (e.g., 5000 PfSPZ per 50 microliter (mcL) dose), Group b: 10,000 PfSPZ in 8 divided doses (e.g., 1250 PfSPZ per 50 mcL dose). Cohort 2: Medium dose, Low Aliquot: Group c: 10,000 PfSPZ in 2 divided doses (e.g., 5000 PfSPZ per 10 mcL dose), Group d: 10,000 PfSPZ in 8 divided doses (e.g., 1250 PfSPZ per 10 mcL dose), Cohort 3: High Dose, Low Aliquot; Group e: 50,000 PfSPZ in 2 divided doses (e.g., 25,000 PfSPZ per 10 mcL dose), Group f: 50,000 PfSPZ in 8 divided doses (e.g., 6,250 PfSPZ per 10 mcL dose)
Drug: Chloroquine — Rescue therapy after challenge: 1500 mg chloroquine base orally, over 48 hours (600 mg at time 0 followed by 300 mg oral base at hours 6, 24 and 48)

SUMMARY:
This study will randomize 30 healthy adult participants to one of three cohorts comprised of six groups of 5 individuals per group to simultaneously receive PfSPZ Challenge via the ID route. The goal will be to determine the optimal dose required to achieve 100% infectivity (ID100) of adult volunteers with P. falciparum malaria.

DETAILED DESCRIPTION:
Study Phase and Design Phase I with experimental malaria challenge. The study will enroll 30 healthy adult participants randomized to one of three cohorts comprised of six groups of 5 individuals per group to simultaneously receive PfSPZ Challenge via the ID route. The goal will be to determine the optimal dose required to achieve 100% infectivity (ID100) of adult volunteers. The parameters of 1) dose (number of sporozoites) 2) number of injections and 3) aliquot volume will be studied; adding to previous data collected at the University of Nijmegen. The following single time point inoculation regimens (a-f) will be assessed: Cohort 1: Medium dose, medium aliquot volume: a. 10,000 PfSPZ ID in 2 divided doses of 50 microliter aliquot volume b. 10,000 PfSPZ ID in 8 divided doses of 50 microliter aliquot volume Cohort 2: Medium dose, low aliquot volume: c. 10,000 PfSPZ ID in 2 divided doses of 10 microliter aliquot volume d. 10,000 PfSPZ ID in 8 divided doses of 10 ml aliquot volume Cohort 3: High dose, low aliquot volume: e. 50,000 PfSPZ ID in 2 divided doses of 10 ml aliquot volume f. 50,000 PfSPZ ID in 8 divided doses of 10 ml aliquot volume. Safety, tolerability and efficacy of the inoculation regimens will be evaluated. All 30 volunteers will be evaluated as part of an inpatient stay (Days 8-18 post-injection) to diagnose and treat Pf malaria infection with chloroquine. Following review, and with the assistance of an independent SMC, 2 regimens will be chosen for further testing in DMID 11-0042. The following criteria strategy will be employed in the order listed: 1. Regimen necessary to achieve ID100 of adult volunteers; 2. Regimen eliciting Pf patency and parasite density (as detected by qRT-PCR) that most closely approximates patency rates experienced after mosquito challenge; 3. Regimen requiring the least number of injections; 4. Regimen utilizing the fewest number of PfSPZ; 5. Volume of administration considered to be the easiest to administer by the clinicians. Chloroquine sub-study: Eighteen of thirty participants (3 volunteers from each of the six groups comprised of 5-subjects/group) will be assigned to participate in a CQ and possibly desethylchloroquine blood and urine study designed to assess the drug kinetics of CQ over the course of four weeks after standard CQ dose administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant female between the ages of 18 and 45 years, inclusive.
2. Women who are not surgically sterile (no history of bilateral tubal ligation, bilateral salpingo-oophorectomy, or hysterectomy), post-menopausal (1 year without menses) or determined otherwise by medical evaluation to be sterile must agree to practice adequate contraception (such as double barrier methods (condoms plus foam or spermicide, diaphragm plus foam or spermicide), licensed intrauterine devices (IUDs), intravaginal or intra/transdermal or oral hormonal methods initiated at least 1 month prior to inoculation or challenge, documented surgical sterilization via tubal ligation the essure procedure or hysterectomy, abstinence or a vasectomized partner). The contraceptive method should remain unchanged throughout the entire study period (56 days). Serologic pregnancy tests will be conducted upon screening. Urine testing will be done on the day of malaria challenge, on the day of the first positive malaria smear and at the conclusion of active surveillance (Day 56).
3. Is in good health, as determined by vital signs (heart rate, blood pressure, oral temperature), medical history, screening 12-lead ECG and a physical examination.
4. Has normal laboratory values (Urinalysis (assessing blood, and protein presence as greater than trace by dipstick), hemoglobin, WBC, platelet count, AST, ALT, bilirubin, glucose, and creatinine) prior to challenge study. Any abnormal screening value for any screening test listed in Table 8 will exclude the participant from the study with the exception of elevated fasting glucose and hematuria >1+ detected during menses for females. Elevated fasting glucose may need to be repeated due to recent carbohydrate consumption and is therefore not a true fasting glucose. Subsequent repeat fasting glucose testing that is in the normal range will be acceptable for participation. For females who are menstruating, urinalysis frequently tests positive for blood and is not an indicator of poor health status or increased risk. This can be repeated if clinically warranted.
5. Able to understand and comply with planned study procedures including an inpatient stay from Day 8-18 after malaria challenge.
6. Provides informed consent prior to any study procedures, correctly answers > 70% on the post consent quiz and is available for all study visits.
7. Willing to avoid non-study related blood donation for 3 years

Exclusion Criteria:

While not a formal exclusion criterion, the deltoid area of both arms will be assessed for marks, burns and other skin damage. If, in the Investigator's opinion, assessment of local reactions could be impaired, the subject may be excluded under criterion 23.

1. Has any known history of malaria infection, is a long-term resident (> 5 years) of a malaria-endemic area, was born and resided in a malaria-endemic area, or has traveled to a malaria-endemic area within the previous 6 months.
2. Has a positive urine pregnancy test prior to malaria challenge (if female of childbearing potential), is lactating, or has the intention to become pregnant within 2 months after enrollment in this study.
3. Use of any antibiotic (that has known or potential antimalarial properties) or antimalarial drug beginning 28 days prior to the screening and extending to Day 56 of study surveillance.
4. Has evidence of increased cardiovascular disease risk (defined as > 10%, 5 year risk) as determined by the method of Gaziano. Risk factors include sex, age (years), systolic blood pressure (mm Hg), smoking staus (current vs. past or never), BMI (kg/mm2), reported diabetes status (yes/no), current treatment for raised blood pressure (yes/no).
5. Is immunosuppressed (e.g., poorly-controlled diabetes mellitus, cirrhosis, renal insufficiency, active malignancy, connective tissue disease, organ transplant) as a result of an underlying illness or treatment.
6. An abnormal ECG, defined as one showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block.
7. Has an active neoplastic disease (excluding nonmelanotic skin cancer) or neoplastic disease within the past 5 years or any history of hematologic malignancy.
8. Is using or intends to continue using oral or parenteral steroids, high-dose inhaled steroids (>800 micrograms/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs (an exception includes asthma for which any oral or inhaled steroid intake will mean exclusion from study enrollment).
9. Has a known history of human immunodeficiency virus, hepatitis B surface antigen positivity, or Hepatitis C infection.
10. Has a history of alcohol or drug abuse in the last 5 years.
11. Has a history of receiving blood products within the 3 months prior to enrollment in this study.
12. Has a history of psoriasis or porphyria, which may be exacerbated after treatment with chloroquine.
13. Has an acute or chronic medical condition that, in the opinion of the investigator, would render malaria challenge unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known liver disease, renal disease, neurological disorders, visual field defects, cardiac disorders, pulmonary disorders, auditory damage, diabetes mellitus, and transplant recipients).
14. Has a history of anaphylactic response to mosquito bites or known allergy to chloroquine, 4-aminoquinoline derivatives, atovaquone/proguanil, (Malarone®), ibuprofen, or acetaminophen that may be used to treat volunteers developing malaria after P. falciparum challenge.
15. Is using or intends to continue using a medication known to cause drug reactions with chloroquine or Malarone®, such as cimetidine, metoclopramide, antacids or kaolin (antacids and kaolin can be administered at least 4 hours from intake of chloroquine).
16. History of retinal or visual field changes, auditory damage, or seizures.
17. History of splenectomy
18. Has known sickle cell trait or laboratory evidence of sickle cell trait.
19. Has an acute illness, including an oral temperature greater than 100.4 degrees F, within 24 hours prior to CHMI.
20. Plans to undergo surgery (elective or otherwise) between enrollment and 4 weeks (28 days) post-challenge
21. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during the 2-month post-challenge period.
22. Has a diagnosis of schizophrenia, bi-polar disease or other major psychiatric condition that makes study compliance difficult (e.g. subjects with psychoses or history of suicide attempt or gesture in the 3 years before study entry, ongoing risk for suicide)
23. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of a positive malaria smear after the malaria challenge during a 56-day surveillance period and stratified by group. | Days 0, 5-18, 20, 22, 24, 26, 28, 35, 42, and 56 .
The number of serious adverse events throughout the duration of the study. | Day 0 to1 year.
The number and severity of solicited systemic symptoms for 14 days following ID administration of PfSPZ. | Within 14 days after PfSPZ administration.
The number and severity of injection site reactions within 14 days following ID administration of PfSPZ. | Within 14 days after PfSPZ administration.
The number and severity of unsolicited adverse events after the malaria challenge during a 56-day surveillance period (day of challenge and 55 subsequent days) but not related to malaria event symptoms. | Days 0-56.

SECONDARY OUTCOMES:
T cell responses, effector/central memory populations, and intracellular cytokine secretion (ICS) against the malaria antigens by Multiparameter Flow Cytometry | Days 0, 5, 14 and 28
Occurrence of a positive real-time quantitative polymerase chain reaction (PCR) after the malaria challenge during a 56-day surveillance period. | Days 0, 5-18, 20, 22, 24, 26, 28, 35, 42, and 56.
Antibody titers to the pre-erythrocytic stage antigens, and by indirect fluorescent antibody test for antibodies to P. falciparum sporozoites, late liver stage parasites, asexual and sexual erythrocytic stages. | Days 0, 5, 14 and 28

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Lyke KE, Laurens MB, Strauss K, Adams M, Billingsley PF, James E, Manoj A, Chakravarty S, Plowe CV, Li ML, Ruben A, Edelman R, Green M, Dube TJ, Sim BKL, Hoffman SL. Optimizing Intradermal Administration of Cryopreserved Plasmodium falciparum Sporozoites in Controlled Human Malaria Infection. Am J Trop Med Hyg. 2015 Dec;93(6):1274-1284. doi: 10.4269/ajtmh.15-0341. Epub 2015 Sep 28. PMID 26416102